CLINICAL TRIAL: NCT04452630
Title: The CardioPostCovid Study: Cardiovascular Consequences After COVID-19
Brief Title: Cardiovascular Consequences After COVID-19
Status: Terminated | Type: Observational
Why Stopped: The study was stopped because the recruitment goal could not be reached.
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-36
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Cardiovascular Consequences After an Episode of COVID 19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid 19 Patients: patients having presented an episode of Covid-19 diagnosed by at least one positive nasopharyngeal RT-PCR test for SARS-Cov-2 and considered recovered.
  Interventions: Other: Infectious Disease and Cardiology Clinical Consultations

INTERVENTIONS:
Other: Infectious Disease and Cardiology Clinical Consultations — Infectious Diseases and Cardiology Clinical Consultations at 1 month and 12 months of recovery from an episode of Covid-19

SUMMARY:
The occurrence of cardiovascular complications in SARS-CoV-2 infections appears to be more frequent than in other viral respiratory infections, probably due to a singular pathophysiology of this coronavirus.

The lack of characterization of cardiovascular damages linked to Covid-19 could have medium and long-term consequences on the prognosis of patients. This problematic could lead to a second major public health problem linked to Covid-19 and it is therefore crucial to keep monitoring and screening patients at risk.

In this context of emerging infectious diseases, of poorly characterized cardiovascular damages during infection and of absence of data on the long-term evolution of the infection, the investigators propose to carry out a prospective and observational cohort study focused on the evaluation and the systematic cardiovascular follow up of patients who survived an episode of Covid-19, regardless of their cardiovascular profiles.

ELIGIBILITY:
Inclusion Criteria:

• All adults affiliated to social security attending the post-Covid follow-up consultation, having presented an episode of Covid-19 diagnosed by at least one positive nasopharyngeal RT-PCR test for SARS-Cov-2 and considered recovered.

Exclusion Criteria:

* Age <18 years old
* Major under guardianship or curatorship
* Absence of non-opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients can be enrolled in this study if they survived to an episode of Covid-19, whether they were hospitalized or not. They must have been diagnosed Covid19 positive according to international recommendations between January 24, 2020 (date of the first case declared in mainland France) and June 30, 2020. They will be offered to participate to the study during the systematic consultations set up at the Nord Hospital for follow-up patients who have been infected.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Presence of at least one clinical, biological and/or imaging cardiovascular anomaly within 1 month of recovering | 1 month
  Describe clinical, biological and imaging cardiovascular data 1 month after recovery from an episode of Covid-19

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No